CLINICAL TRIAL: NCT05509764
Title: Evaluation of Oxygen Threapy by Lung Ultrasound and Oxygen Reserve Index in Patients Undergoing Cesarean Section Under Spinal Anesthesia
Brief Title: The Effect of Oxygen Therapy on Atelectasis
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Manolya ALKAN CANITEZ, Anesthesiologist, Zonguldak Bulent Ecevit University
Other Study IDs: 2021/02
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Atelectasis; Cesarean Section; Hypotension
Keywords: Atelectasis; lung ultrasound; oxygen reserve index; cesarean section
MeSH Terms: conditions — Pulmonary Atelectasis; Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 0: control group
  Interventions: Diagnostic Test: lung ultrasound score
- group 3: 3 Lt/min Oxygen therapy via nasal cannula
  Interventions: Diagnostic Test: lung ultrasound score
- group 6: 6 Lt/min Oxygen therapy via Simple face mask
  Interventions: Diagnostic Test: lung ultrasound score

INTERVENTIONS:
Diagnostic Test: lung ultrasound score — determination of atelectasis by lung ultrasound score

SUMMARY:
In pregnancy, cephalal shift of the diaphragm caused by the enlarged uterus reduces the functional residual capacity and may increase the closure volume and predispose the pregnant woman to airway closure, leading to atelectasis. The development of atelectasis due to dermatomes retained in spinal anesthesia and intraoperative supine position may increase further. Oxygen therapy to be applied may also lead to absorption atelectasis by causing hyperoxia. The aim of our study is to evaluate the effect of oxygen support on the lungs in cesarean section operations under spinal anesthesia by lung ultrasound score and oxygen reserve index.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* ASA I-II
* Patients scheduled for elective cesarean section under spinal anesthesia

Exclusion Criteria:

* alcohol or drug addiction, chronic obstructive pulmonary disease, cardiovascular disease, smokers anemia, liver or kidney disease, coagulation disorders allergic to anesthetic agents, sepsis or bacterial infection, body temperature is below 35°C and above 38°C Multiple pregnancy Preoperative hypoxemia SpO2<94% Diabetes mellitus Hypertension Placenta previa Premature rupture of membranes Intrauterine growth retardation Preeclampsia-eclampsia-fetal distress Polyhydramnios Morbid obesity BMI>45

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — parturients who underwent cesarean section under spinal anesthesia
Study Population: parturients who underwent cesarean section under spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
atelectasis | during the surgery
  measuring atelectasis due to oxygen therapy

SECONDARY OUTCOMES:
APGAR score | 1st and 5th min after delivery
  baby status after delivery
hypotension | during surgery
  maternal hypotension

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Manolya Alkan, Zonguldak, Kozlu
  - Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu

IPD SHARING:
Plan to Share IPD: Yes